CLINICAL TRIAL: NCT04625673
Title: Phase 2, Randomized Study of the Tolerability and Safety of the OsciPulse Device for the Prevention of VTE
Brief Title: OsciPulse Device for the Prevention of VTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: OsciFlex LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 844294; OSC-VTE-001 (Other: University of Pennsylvania)
Record Dates: First submitted 2020-10-27; First posted 2020-11-12 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Thromboembolisms
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Two part, open-label, randomized, crossover study. Part 1 will enroll 3 healthy subjects. Part two will enroll 15-20 in-patient subjects. Part two will have two arms.
  Arm A will wear the OsciPulse then wear the standard IPC device. Arm B will wear the standard IPC device then wear the OsciPulse device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Group A (Active Comparator): Group A will wear the OsciPulse device for the first 3 hours then switch to the standard IPC device for the second 3 hours.
  Interventions: Device: OsciPulse
- Group B (Active Comparator): Group B will wear the standard IPC device for the first 3 hours then switch to the OsciPulse device for the second 3 hours.
  Interventions: Device: OsciPulse

INTERVENTIONS:
Device: OsciPulse — OsciPulse device and standard IPC device
  Other Names: Standard IPC device

SUMMARY:
This is a Phase 2 safety and tolerability trial that will take place in two parts. Part one of the trial will determine the tolerability of the OsciPulse device on healthy subjects who wear the device for up to three hours. Healthy volunteers will answer questionnaires and may undergo an ultrasound test at the end of their participation in the trial.

Part two of the trial will determine the safety and tolerability of the OsciPulse device on subjects admitted to Penn Presbyterian Medical Center. Eligible subjects will be enrolled for 6 hours. In the first 3 hours, subjects will wear the standard of care intermittent pneumatic compression device or the OsciPulse device. In the second 3 hours, the subject's device will be switched and subjects will wear the alternate device not used in the first 3 hours. Subjects will answer questionnaires and may undergo an ultrasound at the end of the first 3 hours and at the end of the second 3 hours (at hour 6).

ELIGIBILITY:
Inclusion Criteria:

Part 1: Adult over the age of 40, generally healthy without a current foot or ankle injury, no history of diagnosed vascular disease including DVT, PE, VTE, post-phlebetic syndrome, or chronic venous insufficiency, mentally alert and understand English proficiently, able to give informed consent

Part 2: Adult over the age of 18, admitted to the at Penn Presbyterian Medical Center, anticipated decreased level of mobility for at least 6 hours as determined by the clinical team in collaboration with study personnel, mentally alert and understand English proficiently, able to give informed consent.

Exclusion Criteria:

Part 1: injury to the lower limbs, skin breaks, abrasion, or irritation in the area of the limb in contact with the OsciPulse device.

Part 2:

1. Inability or contraindication to applying IPC to both legs such as:

   * Evidence of bone fracture in lower extremities
   * Burns in the lower extremities, lacerations, ulcers, active skin infection or dermatitis, & ischemic limb in the legs at the site of IPC placement
   * Acute ischemia in the lower extremities
   * Severe peripheral vascular disease
   * Amputated foot or leg on one or two sides
   * Compartment syndrome
   * Severe lower extremity edema
2. Subjects anticipated to require surgical intervention within six (6) hours of admission
3. Subjects with history of VTE (DVT or PE)
4. Previous vascular surgery
5. Pregnancy or within 6 weeks of postpartum period
6. Limitation of life support, life expectancy < 7 days or palliative care
7. Admitted to an outside hospital more than 24 hours prior to screening
8. A head-unit is unavailable for the 6 hours or more
9. At the discretion of the attending physician and / or clinical team, the subject's participation in the study is believed not to be in the best interest of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Cuker, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part 1 subjects did NOT go on to Part 2. Part 1 were healthy subjects. Part 2 were patients (not healthy subjects). The study protocol describes the 2 separate groups as "part 1" and "part 2" of the study, which is why this terminology was used.
Groups:
- Part 1: OsciPulse in Healthy Subjects: Testing OsciPulse device in healthy subjects.
- Part 2, Group A, OsciPulse, Then Standard IPC: Subjects in Part 2, Group A will wear the OsciPulse device for the first 3 hours then switch to the standard IPC device for the second 3 hours.
  Subjects who participated in Part 1 of the study did NOT participate in Part 2.
- Part 2, Group B, Standard IPC Device, Then OsciPulse: Part 2, Group B subjects will wear the standard IPC device for the first 3 hours then switch to the OsciPulse device for the second 3 hours.
  Subjects who participated in Part 1 of the study did NOT participate in Part 2.
Period: Overall Study
Arm/Group | Part 1: OsciPulse in Healthy Subjects | Part 2, Group A, OsciPulse, Then Standard IPC | Part 2, Group B, Standard IPC Device, Then OsciPulse
Started | 3 | 9 | 11
Completed | 3 | 9 | 10
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part 1, OsciPulse in Healthy Subjects: Part 1 subjects only
- Part 2, Group A, OsciPulse, Then Standard IPC: Group A will wear the OsciPulse device for the first 3 hours then switch to the standard IPC device for the second 3 hours.
- Part 2, Group B, Standard IPC, Then OsciPulse: Group B will wear the standard IPC device for the first 3 hours then switch to the OsciPulse device for the second 3 hours.
- Total: Total of all reporting groups
Arm/Group | Part 1, OsciPulse in Healthy Subjects | Part 2, Group A, OsciPulse, Then Standard IPC | Part 2, Group B, Standard IPC, Then OsciPulse | Total
Number analyzed (Participants) | 3 | 9 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 7 | 9 | 19
  >=65 years | 0 | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 5 | 13
  Male | 0 | 4 | 6 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 3 | 4 | 5 | 12
  African American | 0 | 4 | 5 | 9
  Asian | 0 | 0 | 1 | 1
  Unknown | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 9 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Part 1 - Subject's Response to Tolerability Questionnaire
Description: Tolerability will be measured by subject's response to questionnaires to assess their experience with the device. This will be measured on a linear 100 mm visual acuity scale measured in millimeters. Subjects are provided with the scale and asked to make a mark on the line that corresponds to their experience with the device. The least favorable rating is on the left hand side, the most favorable rating is on the right hand side of the scale. The mark on the line is measured in millimeters, resulting in least favorable scores having a lower score, and most favorable ratings having a higher score.
Time Frame: up to 3 hours
Population: This outcome measure is applicable to part 1 only.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1, Healthy Subjects: Healthy subjects
Arm/Group | Part 1, Healthy Subjects | Part 2, Group A, OsciPulse, Then Standard IPC | Part 2, Group B, Standard IPC, Then OsciPulse
Number analyzed (Participants) | 3 | 0 | 0
Participants
  No discomfort | 3 | 0 | 0
  Mild discomfort | 0 | 0 | 0
  Significant discomfort | 0 | 0 | 0

2. Primary Outcome: Part 1 - Safety Assessment Through Collection of Adverse Events
Description: Safety will be assessed by collecting & reviewing all adverse events while subject is wearing the device.
  Subjects will indicate if the device caused 1) no discomfort, 2) mild discomfort, or 3) significant discomfort. To move on to Part 2, all subjects in Part 1 must indicate that there was not "significant discomfort."
Time Frame: up to 3 hours
Population: This outcome measure is applicable to part 1 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Healthy Subjects | Part 2, Group A, OsciPulse, Then Standard IPC | Part 2, Group B, Standard IPC, Then OsciPulse
Number analyzed (Participants) | 3 | 0 | 0
Participants | 0 | 0 | 0

3. Primary Outcome: Part 2 - Subject's Response to Tolerability Questionnaire
Description: Tolerability will be measured by subject's response to questionnaires to assess their experience with the device. This will be measured on a linear 100mm visual acuity scale measured in millimeters. Subjects are provided with the scale and asked to make a mark on the line that corresponds to their experience with the device. The minimum (least favorable) rating is on the left hand side and is equal to zero (0), the maximum (most favorable) rating is on the right hand side of the scale and is equal to one hundred (100). For Comfort, scores range from "very disruptive" (0) to "no effect" (10). For Disruption, scores range from "very disruptive" (0) to "no effect" (10). For Noise, scores range from "very loud" (0) to "not noticeable" (10). For Movement, scores range from "very restrictive" (0) to "no effect" (10). The mark on the line is measured in millimeters, resulting in minimum (least favorable) scores having a lower score, and maximum (most favorable) ratings having a higher score.
Time Frame: 6 hours
Population: This outcome measure is applicable to part 2 only, which had groups A and B.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Part 2, Group A, OsciPulse, Then Standard IPC | Part 2, Group B, Standard IPC, Then OsciPulse
Number analyzed (Participants) | 6 | 6
score on a scale
  Comfort-OsciPulse | 7.2 [0 to 10] | 6.08 [0 to 10]
  Comfort-Standard IPC | 6.8 [0 to 10] | 9.03 [0 to 10]
  Disruption-OsciPulse | 7 [0 to 10] | 4.47 [0 to 10]
  Disruption-Standard IPC | 7.48 [0 to 10] | 8.18 [0 to 10]
  Noise-OsciPulse | 3.48 [0 to 10] | 4.08 [0 to 10]
  Noise-Standard IPC | 7.6 [0 to 10] | 7.05 [0 to 10]
  Movement Interference-OsciPulse | 5.6 [0 to 10] | 7.15 [0 to 10]
  Movement Interference-Standard IPC | 4.78 [0 to 10] | 6.7 [0 to 10]

4. Primary Outcome: Part 2 - Safety Assessment Through Collection of Adverse Events.
Description: Safety will be assessed by collecting all adverse events while the subject is wearing the device.
Time Frame: 6 hours
Population: This outcome measure is applicable to part 2 only, which had groups A and B.
  The subject consented to Part 2, Group B had an AE prior to being able to use either device. So subject was consented to study but did not have an AE with either standard or investigational device.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2, Group A, OsciPulse, Then Standard IPC: Group A will wear the OsciPulse device for the first 3 hours then switch to the standard IPC device for the second 3 hours.
  Subjects who participated in Part 1 of the study did NOT participate in Part 2.
- Part 2, Group B, Standard IPC, Then OsciPulse: Group B will wear the standard IPC device for the first 3 hours then switch to the OsciPulse device for the second 3 hours.
  Subjects who participated in Part 1 of the study did NOT participate in Part 2.
  One subject consented but did not participate in the study.
Arm/Group | Part 2, Group A, OsciPulse, Then Standard IPC | Part 2, Group B, Standard IPC, Then OsciPulse
Number analyzed (Participants) | 9 | 11
Participants
  No AEs-OsciPulse | 9 | 10
  No AEs-Standard IPC | 9 | 10
  AEs-OsciPulse | 0 | 0
  AEs-Standard IPC | 0 | 0
  AEs-not related to device | 0 | 1

ADVERSE EVENTS:
Time Frame: 6 hours
Description: One subject was removed from study due to SAE before inv. product was administered. This subject is included in the safety assessment only. Subjects who participated in Part 1 did NOT go on to Part 2.
Groups:
- Part 1: Healthy Subjects: OsciPulse in Healthy Subjects
- OsciPulse: Those wearing the OsciPulse device.
- Standard IPC: Those wearing the standard IPC device.
Arm/Group | Part 1: Healthy Subjects | OsciPulse | Standard IPC
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 0/3 | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Healthy Subjects (N=3) | OsciPulse (N=20) | Standard IPC (N=20)
Pancreatitis (Gastrointestinal disorders) | NA | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT04625673/Prot_SAP_000.pdf